CLINICAL TRIAL: NCT03530150
Title: Pirfenidone and Its Efficacy in Wound Re-Epithelization in Patients With Second-Degree Burns: A Proof-of-Concept Randomized Controlled Trial
Brief Title: Pirfenidone and Its Role in Burn Wound Healing
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, Gabriel Angel Mecott-Rivera, Principal Investigator, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CP14-004
Record Dates: First submitted 2018-05-07; First posted 2018-05-21 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Second-degree Burn
Keywords: Burns; Partial-thickness burn wounds; Re-epithelization; Second-Degree Wound; Pirfenidone; Wound Healing
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: Burn patients will be divided to receive either 600 mg of pirfenidone or usual care
Who Masked: Investigator, Outcomes Assessor
Masking Description: The principal investigator, the person in charge of gathering the data, and the person analyzing the data will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pirfenidone 600 mg (Active Comparator): Burn patients randomly allocated to this group will receive pirfenidone 600 mg orally once per day for 21 days additionally to the coverage of the wound with non-adherent gauzes and bandages. The aforementioned coverings will be changed every 3 or 4 days until a complete re-epithelization is achieved.
  Interventions: Drug: Pirfenidone Oral Product
- Usual Care (No Intervention): Burn patients randomly allocated to this group will only be treated by the usual care of our hospital which consists in covering the wound with non-adherent gauzes and bandages. These covering will be changed every 3 or 4 days until a complete re-epithelization is achieved.

INTERVENTIONS:
Drug: Pirfenidone Oral Product — A pill containing 600 mg of pirfenidone
  Other Names: Kitoscell
  Arms: Pirfenidone 600 mg

SUMMARY:
Burn patients which skin has been lost a rapid growth of the skin is a foremost in their treatment. Due to the injury, burn patients undergo a systemic inflammation that helps the skin heal faster. However, several studies have shown that this inflammation increases the levels of several inflammatory molecules that impairs skin growing, which further delays the recovery of burn patients. As such, by inhibiting these inflammatory molecules with the administration of a medication called pirfenidone burn patients might present faster rates of skin growth and recovery. Thus, patients suffering from a burn injury will be recruited at the emergency department of the Hospital University in Monterrey Mexico. Afterward, patients will be randomized to either receive pirfenidone 600 mg orally once per day or usual care consisting of covering the wound with hydrocolloid dressings. To assess the amount of newly growth skin investigators will take a small piece of the skin to further evaluate it through a microscope.

ELIGIBILITY:
Inclusion Criteria:

* Patients with second-degree burns from any etiology with less than 24 hours of evolution.

Exclusion Criteria:

* Patients <18 years old
* Patients allergic to pirfenidone
* Pregnant patients
* Patients with renal or hepatic failure
* Patients who are not able to take the medication orally
* Conditions or drugs that alter wound healing (i.e. any kind of diabetes, lupus, having a history of using steroids, rheumatoid arthritis)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-06-22 (Actual); Study Completion 2017-06-22 (Actual)

PRIMARY OUTCOMES:
Epidermal re-epithelization | Day 7
  Thickness of the epidermal re-epithelization measured in micrometers using a digitial image software

SECONDARY OUTCOMES:
Presence of Fibrosis | Day 0 and 7
  A qualitative assessment of the presence of fibrotic tissue in the extracellular matrix using a light field microscope.
Basal Membrane Integrity | Day 0 and 7
  A qualitative assessment of the presence and integrity of the basal membrane using a light field microscope.
Presence of Collagen Fibers | Day 0 and 7
  A qualitative assessment of the presence of collagen fibers in the dermis using a light field microscope.
Clinical Evaluations of Wound's Re-Epithelization | Day 7
  Clinical evaluation of wound's re-epithelization based on the judgement of an experienced plastic surgeon

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel A Mecott-Rivera, MMS, Principal Investigator — Universidad Autonoma de Nuevo Leon

IPD SHARING:
Plan to Share IPD: Yes
All information will be delivered by request.
  Possible individual participant data includes:
  Database Original Protocol Informed Consent
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available from May 2018 to May 2020